CLINICAL TRIAL: NCT00322231
Title: A Phase III Clinical Trial to Study the Safety, Tolerability and Immunogenicity of Zoster Vaccine Live in Subjects With a History of Herpes Zoster
Brief Title: A Study of an Investigational Zoster Vaccine, in Subjects With a History of Herpes Zoster (V211-014)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: V211-014; 2006_010
Record Dates: First submitted 2006-05-02; First posted 2006-05-05 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ZOSTAVAX™ / Placebo (Experimental): Zoster vaccine live on Day 1 (Period 1), placebo on Week 4 (Period 2)
  Interventions: Biological: zoster vaccine live (ZOSTAVAX™); Biological: Comparator: Placebo
- Placebo / ZOSTAVAX™ (Experimental): Placebo on Day 1 (Period 1), zoster vaccine live on Week 4 (Period 2)
  Interventions: Biological: zoster vaccine live (ZOSTAVAX™); Biological: Comparator: Placebo

INTERVENTIONS:
Biological: zoster vaccine live (ZOSTAVAX™) — 1 dose 0.65 mL/dose subcutaneous injection of zoster vaccine live
  Other Names: Zostavax
Biological: Comparator: Placebo — 1 dose 0.65 mL/dose subcutaneous injection of placebo.

SUMMARY:
The purpose of this study is to determine whether the investigational zoster vaccine, is generally well tolerated when administered to participants with a history of herpes zoster.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 50 years of age with a history of herpes zoster ≥ 5 years prior to enrollment

Exclusion Criteria:

* History of allergy to any vaccine component
* Prior receipt of a varicella or zoster vaccine
* Ability to defend against infection is suppressed by a medical condition or medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Mills R, Tyring SK, Levin MJ, Parrino J, Li X, Coll KE, Stek JE, Schlienger K, Chan IS, Silber JL. Safety, tolerability, and immunogenicity of zoster vaccine in subjects with a history of herpes zoster. Vaccine. 2010 Jun 7;28(25):4204-9. doi: 10.1016/j.vaccine.2010.04.003. Epub 2010 Apr 21. PMID 20416263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 9 sites in the United States.
  First patient enrolled: May-2006; Last patient last visit: July - 2007
Groups:
- ZOSTAVAX™ / Placebo: 0.65mL of Zoster vaccine live injected subcutaneously on Day 1 (Period 1) followed by 0.65mL of placebo injected subcutaneously at Week 4 (Period 2)
- Placebo / ZOSTAVAX™: 0.65mL of placebo injected subcutaneously on Day 1 (Period 1) followed by 0.65mL of Zoster vaccine live injected subcutaneously at Week 4 (Period 2)
Period: Period 1
Arm/Group | ZOSTAVAX™ / Placebo | Placebo / ZOSTAVAX™
Started | 51 | 50
Completed | 51 | 50
Not Completed | 0 | 0
Period: Period 2
Arm/Group | ZOSTAVAX™ / Placebo | Placebo / ZOSTAVAX™
Started | 51 | 49 (One participant was lost between Period 1 and Period 2)
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX™ / Placebo | Placebo / ZOSTAVAX™ | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Customized [Number; unit: participants]
  50 to 59 Years of age | 10 | 10 | 20
  ≥ 60 Years of age | 41 | 40 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 24 | 60
  Male | 15 | 26 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 4
  Black | 3 | 3 | 6
  Hispanic American | 0 | 2 | 2
  White | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Vaccine-related Serious Adverse Experiences (SAEs) for 28 Days Postvaccination
Description: SAEs are AEs at any dose that: Results in death or persistent/significant disability/incapacity; or prolongs an existing inpatient hospitalization or Is life threatening; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose or Is an other important medical event
Time Frame: To Day 28 postvaccination
Population: All vaccinated participants were evaluated for safety. This was a crossover study. All participants received one dose each of ZOSTAVAX™ and placebo. Data below reflect SAEs reported after receipt of ZOSTAVAX™ or placebo.
Measure: Number; unit: Participants
Groups:
- ZOSTAVAX™: Participants who received ZOSTAVAX™ in the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™ group (see participant flow section) are included
- Placebo: Participants who received placebo in the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™ Group (see participant flow section) are included.
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 100 | 101
Participants
  With Vaccine-related SAEs | 0 | 0
  Without Vaccine-related SAEs | 100 | 101

2. Secondary Outcome: Geometric Mean Titer (GMT) of Varicella-zoster Virus (VZV) Antibody Responses at 4 Weeks Postvaccination
Description: The GMT of the VZV-specific antibody responses as measured by gpELISA (glycoprotein enzyme-linked immunosorbent assay) at the prespecified day ranges at prevaccination and 4 weeks postvaccination
Time Frame: 4 weeks postvaccination
Population: Per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Groups:
- ZOSTAVAX™: Participants who received ZOSTAVAX™ in both, the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™ group (see participant flow section) are included.
- Placebo: Participants who received placebo (at Day 1) in Placebo / ZOSTAVAX™ group. Participants who received ZOSTAVAX™ at (Day 1) in the ZOSTAVAX™ / Placebo group were excluded to avoid a possible carry-over effect of ZOSTAVAX™ on immunogenicity measurements.
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 100 | 50
gpELISA units/mL | 810.1 [688.3 to 953.4] | 391.1 [291.9 to 523.9]

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titers From Prevaccination to 4 Weeks Postvaccination
Description: GMFR of the VZV antibody response at the prespecified day ranges prevaccination and 4 weeks postvaccination
Time Frame: From prevaccination (baseline) to 4 weeks postvaccination
Population: Per-protocol population
Measure: Number (95% Confidence Interval); unit: Geometric mean fold rise
Groups:
- ZOSTAVAX™: Participants who received ZOSTAVAX™ in both, the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™ group are included. In addition, 5 participants from the Placebo / ZOSTAVAX™ group were excluded in the prevaccination summaries (since their specimens were damaged or collected out of day range), and are not in the analysis.
- Placebo: Participants included in this analysis were those who received Placebo in Placebo /ZOSTAVAX™ group (on Day 1). Participants who received ZOSTAVAX™ in the ZOSTAVAX™ / Placebo group were excluded in order to avoid a possible carry-over effect of ZOSTAVAX™ on immunogenicity measurements. In addition, 5 participants from the Placebo / ZOSTAVAX™ group were excluded in the prevaccination summaries (since their specimens were damaged or collected out of day range), and are not in the analysis.
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 95 | 45
Geometric mean fold rise | 2.1 [1.8 to 2.4] | 1.0 [0.9 to 1.1]

ADVERSE EVENTS:
Time Frame: Day 1 - 28 following each vaccination
Description: Injection-site adverse experiences (AEs), rashes, oral temperatures (if the participant felt febrile), and other AEs were recorded by the participant on a Vaccination Report Card which was reviewed by the study site personnel at the end of each 28-day follow-up period.
  The participants at risk are ITT population with follow-up.
Groups:
- ZOSTAVAX™: All participants that received ZOSTAVAX™ from both, the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™ group. Two participants that received ZOSTAVAX™ were lost to follow up and not included in the analysis.
- Placebo: All participants that received Placebo in both, the ZOSTAVAX™ / Placebo group and the Placebo / ZOSTAVAX™. Five participants that received placebo were lost to follow up and not included in the analysis.
Arm/Group | ZOSTAVAX™ | Placebo
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/96
Other Adverse Events (participants affected / at risk) | 45/98 | 4/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX™ (N=98) | Placebo (N=96)
Injection Site Erythema (General disorders) | 33 | 3
Injection Site Pain (General disorders) | 36 | 1
Injection Site Pruritus (General disorders) | 5 | 0
Injection Site Swelling (General disorders) | 26 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.